CLINICAL TRIAL: NCT03332576
Title: Phase 1b Study of Extended Dosing of an Immunotherapeutic Vaccine, DPX-Survivac With Low Dose Cyclophosphamide in Patients With Surgically Operable or Advanced Stage Ovarian, Fallopian Tube or Peritoneal Cancer.
Brief Title: Phase 1b Study of a Cancer Vaccine to Treat Patients With Advanced Stage Ovarian, Fallopian or Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoVaccine Technologies, Inc. (IMV Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-DPX-Survivac-03
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: vaccine; immunotherapy; combination therapy
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): 6 Doses DPX-Survivac (2 prime q3w, 4 boost q8w)
  Low dose cyclophosphamide
  Interventions: Biological: DPX-Survivac; Drug: Cyclophosphamide
- Cohort 2 (Experimental): 6 Doses DPX-Survivac (2 prime q3w, 4 boost q8w)
  Low dose cyclophosphamide
  Interventions: Biological: DPX-Survivac; Drug: Cyclophosphamide
- Cohort 3 (Experimental): 3 Doses DPX-Survivac (1 prime, 2 boost q8w)
  Low dose cyclophosphamide
  Interventions: Biological: DPX-Survivac; Drug: Cyclophosphamide
- Cohort 4 (Experimental): 5 Doses DPX-Survivac (2 prime q6w, 3 boost q6w)
  Low dose cyclophosphamide
  Interventions: Biological: DPX-Survivac; Drug: Cyclophosphamide
- Cohort 5 (Experimental): 5 Doses DPX-Survivac/DPX-Survivac(Aqueous) (2 prime q4w, 3 boost q4w)
  Low dose cyclophosphamide
  Interventions: Biological: DPX-Survivac; Biological: DPX-Survivac(Aqueous); Drug: Cyclophosphamide

INTERVENTIONS:
Biological: DPX-Survivac — SubQ injection
Biological: DPX-Survivac(Aqueous) — SubQ injection
  Arms: Cohort 5
Drug: Cyclophosphamide — PO BID

SUMMARY:
As a follow-on study to NCT01416038, this study is designed to identify the optimal dosage of immunotherapeutic survivin vaccine DPX-Survivac and low dose oral cyclophosphamide. The combination treatment is being evaluated in a non-randomized, multi-cohort study as post-chemotherapy treatment for patients with late-stage ovarian, fallopian tube, or peritoneal cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed stage IIc-IV epithelial ovarian, fallopian tube or peritoneal cancer
* Complete or partial response following standard of care surgery and first line chemotherapy
* May have one disease recurrence with complete or partial response or stable disease following standard of care second line care treatment
* Previous investigational biologic therapy allowed, must be more than 56 days prior to first injection
* Previous treatment with bisphosphonate allowed, must be completed 14 days prior to first injection
* Ambulatory with an ECOG 0-1
* Life expectancy > 6 months
* Meet protocol-specified lab requirements
* Provide informed consent and have ability to comply with protocol requirements

Key Exclusion Criteria:

* Concurrent chemotherapy, radiation therapy, immunotherapy are excluded (washout periods as specified in protocol)
* Prior receipt of survivin based vaccines
* Participation in prior therapeutic adjuvant ovarian cancer studies, except for platinum-based adjuvant studies
* Progressive disease (rising CA-125 acceptable)
* More than one course of chemotherapy for recurrent disease
* Concurrent bevacizumab as maintenance therapy
* Concurrent second malignancy other than non-melanoma skin cancer, cervical carcinoma in situ, or controlled bladder cancer
* History of autoimmune disease
* Recent history of thyroiditis
* Presence of a serious acute infection or chronic infection
* Brain metastases
* Other serious intercurrent chronic or acute illness
* Ongoing treatment with steroid therapy or other immunosuppressive
* Acute or chronic skin disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-08-23 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse event reporting (CTCAE) | up to 11 months

SECONDARY OUTCOMES:
Cell mediated immunity as measured by the antigen specific response in peripheral blood | up to 11 months
Impact on residual tumour | up to 11 months
  Evaluated by standard of care radiology and CA-125

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Winthrop University Hospital, Mineola, New York
  - Lenox Hill Hospital, New York, New York
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No